CLINICAL TRIAL: NCT04085952
Title: Comparing Anterior Prolapse Repair With and Without Allograft Use: A Randomized Control Trial With Long Term Follow-Up
Brief Title: Anterior Prolapse Repair With and Without Graft Augmentation
Acronym: ARCUS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Endeavor Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EH04-302
Record Dates: First submitted 2017-04-28; First posted 2019-09-11 (Actual); Last update posted 2019-09-11 (Actual); Status verified 2019-09

CONDITIONS: Pelvic Organ Prolapse
Keywords: pelvic organ prolapse, vaginal graft
MeSH Terms: conditions — Pelvic Organ Prolapse

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- anterior colporrhaphy with dermal graft (Experimental): Patients randomized to this arm underwent anterior colporrhaphy with dermal graft augmentation (ARUCS) during their surgery for pelvic organ prolapse.
  Interventions: Procedure: dermal graft (ARCUS repliform) for anterior colporrhaphy
- anterior colporrhaphy suture based (Active Comparator): Patients randomized to this arm underwent anterior colporrhaphy with suture based repair (native tissue) during their surgery for pelvic organ prolapse. This is and was the most common practice for anterior colporrhaphy.
  Interventions: Procedure: suture based anterior colporrhaphy

INTERVENTIONS:
Procedure: dermal graft (ARCUS repliform) for anterior colporrhaphy — At the time of surgery patients were randomized to anterior colporrhaphy with dermal graft augmentation
  Arms: anterior colporrhaphy with dermal graft
Procedure: suture based anterior colporrhaphy — At the time of surgery patients were randomized to anterior colporrhaphy with a suture based repair
  Arms: anterior colporrhaphy suture based

SUMMARY:
This is a randomized control trial comparing anterior colporrhaphy with augmentation with dermal allograft (ARCUS) to anterior colporrhaphy with a suture-based repair (native tissue). Patients were randomized to one treatment and then were followed post-operatively for 7-10 years. Prior to surgery patients had a POPQ vaginal prolapse exam and completed a quality of life questionaire (PFDI). They had a repeat POPQ exam and quality of life questionaires at their post-op operative visits. We compare recurrent prolapse rates between these 2 groups.

DETAILED DESCRIPTION:
Objective: To determine whether dermal allograft (ARCUS) reduces anterior prolapse recurrence at 1 and 7-10 years post-operatively. Our central question is whether we can reduce the rate of rate of anterior compartment prolapse recurrence after surgical repair, is the recurrence rate reduced with allograft use, and does this benefit hold up over time?

Methods: Patient will be randomized by computer generated block randomization to native tissue (suture based) anterior colporrhaphy or colporrhaphy with graft (ARCUS) usage. Neither patients nor surgeons will be blinded due to the nature of the surgery. Patients will be followed for 7-10 years post-operatively. Participants will complete a POPQ exam and the PFDI (Pelvic Floor Distress Inventory) questionnaire pre-operatively. Patients will return for a POPQ exam at 1 year post-operatively and complete the PFDI (Pelvic Floor Distress Inventory) and PISQ (Sexual Function for Women with: POP, Urinary Incontinence and/or Fecal Incontinence) questionnaires. Patients will be asked to return to the office for a research visit 7-10 years post-operatively for a POPQ exam and to complete quality of life questionnaires including PFDI 20 (Pelvic floor distress inventory), PISQ-R (Sexual Function for Women with: POP, Urinary Incontinence and/or Fecal Incontinence, Revised), and PGI (Patient global assessment of improvement).

ELIGIBILITY:
Inclusion Criteria: Any patient planning to undergo surgery for anterior compartment prolapse, English speaking.

-

Exclusion Criteria: Any patient who does not speak English due to standardized English language based questionaires, and patients without anterior compartment prolapse.

-

Ages: 18 Years to 100 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2005-01; Primary Completion 2009-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
1-Year Recurrent prolapse- anatomic | 1 year post-operative
  Failure of prolapse surgery as measured by changes in POPQ measurements, Aa and Ba to -1 or greater
7-10 Years Recurrent prolapse-anatomic | 7-10 years post-operative
  Failure of prolapse surgery as measured by changes in POPQ measurements, Aa and Ba to -1 or greater

SECONDARY OUTCOMES:
1 Year composite score | 1 year post-operative
  Failure of prolapse surgery as measured as a composite outcome including anatomic failure measured by changes to Aa and Ba points to -1 or greater, "yes" to PFDI question #3, and retreatment with pessary or surgery for anterior compartment prolapse
7-10 years composite score | 7-10 years post-operative
  Failure of prolapse surgery as measured as a composite outcome including anatomic failure measured by changes to Aa and Ba points to -1 or greater, "yes" to PFDI question #3, and retreatment with pessary or surgery for anterior compartment prolapse

CONTACTS AND LOCATIONS:
Overall Officials: Peter Sand, MD, Principal Investigator — North Shore Research Institute

IPD SHARING:
Plan to Share IPD: No